CLINICAL TRIAL: NCT06517589
Title: Process-based Therapy vs. Routine-CBT for Difficult-to-treat Anxiety Disorders and Depression
Brief Title: Process-based Therapy for Difficult-to-treat Anxiety Disorders and Depression
Acronym: PBTRAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrich Stangier, Director of the Department of Clinical Psychology and Psychotherapy and Center for Psychotherapy, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: III L5-519/05.000.002
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety Disorder
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Process-based Cognitive Behavioral Therapy (Experimental): In PBT (20 sessions), treatment is initiated by a collaborative interpretation of the dynamic network model using smartphone-based Ecological Momentary Assessment collected during the baseline. Based on the outcome of the dynamic network model, interventions are selected on the basis of empirical evidence for mechanisms of change matching to the central node of the individual patient, besides feedback loops and self-loops, as the key process maintaining the maladaptive pattern. Interventions are conceptualized in the evolutionary framework as variation, selection and retention of an adaptive mode of the central node related to the specific context of the problem. The change of this variable is monitored using daily judgements on the basis of EMA. Further treatment planning focuses on additional targets to establish the adaptive modes of the dimensions as defined in the positive network model. Concomitant medication is allowed and will be controlled in statistical analyses.
  Interventions: Other: Process-based Cognitive Behavioral Therapy (PBT)
- Traditional Cognitive Behavioral Therapy (Active Comparator): In r-CBT (20 sessions) a naturalistic setting is retained for treatment decisions. Treatment planning follows traditional theories about the effects of the interventions on factors maintaining the disorder, e.g. avoidance and exposure in anxiety disorder or reduced reinforcement of activities and behavioral activation in depression. Interventions are selected on the basis of common treatment manuals related to diagnoses, e.g. CBT for depression. Individual data from the behavioral analysis are used to taylor the techniques to the problem behaviors or dysfunctional thoughts of patients. Treatment process focuses mainly on the implementation of the manualized interventions adapted to the individual patient as recommended in the National guidelines for treatment of depression and anxiety disorders. Concomitant medication is allowed and will be controlled in statistical analyses.
  Interventions: Other: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Other: Process-based Cognitive Behavioral Therapy (PBT) — PBT (20 sessions), intervention planning based on the use of EMA data, feedback of dynamic network analysis and matching of interventions to central nodes of the network.
  Arms: Process-based Cognitive Behavioral Therapy
Other: Cognitive Behavioral Therapy (CBT) — CBT (20 sessions), intervention planning as usual based on manual.
  Arms: Traditional Cognitive Behavioral Therapy

SUMMARY:
The aim of this study is to test the relative efficacy of Process-based Therapy compared to traditional CBT delivered in routine practice (r-CBT) for difficult-to-treat anxiety disorders and depression.

DETAILED DESCRIPTION:
Process-based Therapy (PBT) is a new framework to intervention planning, based on the use of ecological momentary assessment (EMA) data, feedback of dynamic network analysis and matching of interventions to central nodes of the network. Although preliminary support for its applicability has been reported from a single-case study, there are no data on the feasibility and effectiveness in a larger clinical sample. The investigators have translated a Training Manual of PBT and modified for delivery of CBT in Mental Health Service. The aim of this study is to test the relative efficacy of PBT compared to traditional CBT delivered in routine practice (r-CBT) for difficult-to-treat anxiety disorders and depression.

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-5 diagnosis of depressive or anxiety disorder
* At least two unsuccessful attempts of pharmacological or psychological treatment according to the German guidelines for the treatment of depression or anxiety disorders (Arbeitsgemeinschaft der Wissenschaftlichen Medizinischen Fachgesellschaften, AWMF)
* Age 18-65 years
* Sufficient knowledge of the German language
* Participating patients are not required to discontinue medication, but to keep medication constant over the treatment period

Exclusion Criteria:

* Increased suicidality
* Substance abuse or dependency
* Borderline personality disorder
* Pervasive developmental disorder
* Psychotic disorder
* Eating disorder
* Bipolar disorder
* Severe physical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Emotional distress, minimum value=0, maximum value=63, higher scores mean worse outcome

SECONDARY OUTCOMES:
Euroqol-5D (EQ-5D) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Health related quality of life, minimum health state=11111, maximum health state=55555, higher scores in health state mean worse outcome, minimum health score=0, maximum health score=100, higher scores in health score mean better outcome
Positive-Mental Health Scale (PMH) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Positive mental health, minimum value=9, maximum value=36, higher scores mean better outcome
Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Pleasure in interpersonal situations, minimum value=17, maximum value=102, higher scores mean better outcome
Depression Anxiety Stress Scale (DASS-10) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Psychological symptoms of distress, depressive and anxious symptoms, minimum value=0, maximum value=30, higher scores mean worse outcome
Acceptance and Action Questionnaire Version 2 (AAQ-2) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Psychological flexibility and acceptance, minimum value=7, maximum value=49, higher scores mean worse outcome
Reflective Functioning Questionnaire (RFQ-8) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Reflective Functioning, minimum value=8, maximum value=56, higher scores on the uncertainty dimension mean worse outcome, higher scores in the certainty dimension mean better outcomes
Client Satisfaction Questionnaire (CSQ-8) | Assessed at post-treatment at week 32
  Client Satisfaction, minimum value=8, maximum value=32, higher scores mean better outcome
Process-based Assessment Tool (PBAT) | Assessed at inclusion, at pre-treatment, at post-treatment (week 32) and at 6 month follow-up
  Variation, selection and retention of adaptive behavior, minimum value=0, maximum value=1800, higher scores mean better outcome
Cognitive-Behavioral-Therapy Skills Questionnaire (CBTSQ) | Assessed at inclusion, pre-treatment, weekly during the treatment (from week 11 to 30), at post-treatment (week 32) and at 6 month follow-up
  Patients use of CBT interventions, minimum value=6, maximum value=42, higher scores mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- JWGUniversity, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main publication of outcomes, after deidentification (text, tables, figures, and appendices) will be shared. Further Study Protocol, Analysis Plan, Informed Consent Form and Analytic Code will be shared to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication. Data are available for 5 years at a third party website (Link to be included).
Access Criteria: Proposals should be directed to stangier@psych.uni-frankfurt.de. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Stangier U, Kohl V, Gorg N, Sendig L, Hufschmidt B, Bonarius D, Nemani A, Ebert M, Hofmann SG. Process-based therapy vs. routine-CBT for difficult-to-treat mood and anxiety disorders: study protocol for a randomized controlled trial. Trials. 2024 Dec 19;25(1):838. doi: 10.1186/s13063-024-08689-3. PMID 39702504
- See also: Website — https://www.psychologie.uni-frankfurt.de/137433169/PBTRAND

DOCUMENTS (1):
  • Study Protocol (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT06517589/Prot_001.pdf